CLINICAL TRIAL: NCT01239082
Title: CSP #577 - Colonoscopy vs. Fecal Immunochemical Testing in Reducing Mortality From Colorectal Cancer
Brief Title: Colonoscopy Versus Fecal Immunochemical Test in Reducing Mortality From Colorectal Cancer (CONFIRM)
Acronym: CONFIRM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 577
Record Dates: First submitted 2010-11-09; First posted 2010-11-11 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Other): Colonoscopy (one time screening)
  Interventions: Procedure: Colonoscopy
- Arm 2 (Other): FIT (annually)
  Interventions: Procedure: FIT

INTERVENTIONS:
Procedure: Colonoscopy — One time screening Colonoscopy to screen for colorectal cancer
  Arms: Arm 1
Procedure: FIT — Annual FIT testing
  Arms: Arm 2

SUMMARY:
Colorectal cancer (CRC) is currently the second most common cause of cancer death in the United States, and one of the most preventable cancers. It has been shown in several randomized controlled trials that screening using fecal occult blood testing (FOBT) reduces CRC mortality by 13-33%. While there is strong consensus amongst experts regarding the value of CRC screening, the best approach to screening is not clear. Of the widely recommended modalities, FOBT and colonoscopy are the most commonly used within the United States. FOBT is inexpensive, non-invasive, and its use as a screening tool is supported by the highest quality evidence (i.e. randomized controlled trials). Moreover, newer FOBT, such as fecal immunochemical tests or FITs, have advantages over conventional FOBT in terms of both test characteristics and ease of use that make them quite attractive as a population-based screening tool.

While colonoscopy is invasive and has higher up-front risks and costs than FOBT, it does afford the opportunity to directly assess the colonic mucosa and is widely believed to be the best test to detect colorectal cancer. In addition, colonoscopy allows for the detection and removal of colorectal adenomas -a well recognized colorectal cancer precursor. There is indirect evidence that suggests colonoscopy is effective in reducing colorectal cancer mortality, but to date, no large clinical trials have been completed to support this assumption. While colonoscopy use is increasing, data is emerging that colonoscopy may not be as effective as previously believed. Prior support for colonoscopy as a screening test relied upon effectiveness estimates that now appear to be overly optimistic. Given the invasive nature of colonoscopy, the associated small, but real risk of complications, and dramatically higher costs than other screening tests, it is especially important to determine the true comparative effectiveness of colonoscopy relative to other proven non-invasive options.

The investigators propose to perform a, large, simple, multicenter, randomized, parallel group trial directly comparing screening colonoscopy with annual FIT screening in average risk individuals. The hypothesis is that colonoscopy will be superior to FIT in the prevention of colorectal cancer mortality measured over 10 years. Individuals will be enrolled if they are currently eligible for CRC screening (e.g. no colonoscopy in the past 10 years and no FOBT in the past 1 year) and are between 50 and 75 years of age. The investigators will exclude individuals for whom colonoscopy is indicated (e.g. signs or symptoms of CRC, first degree family member with CRC, personal history of colorectal neoplasia or inflammatory bowel disease).

All participants will complete baseline demographic, medication, and lifestyle questionnaires (e.g. diet, non-steroidal anti-inflammatory use, frequency of exercise) prior to randomization in a 1:1 ratio to either screening colonoscopy or annual FIT screening (Figure 1). Those testing positive by FIT will undergo evaluation to determine appropriateness for colonoscopy. Screening will be performed in a manner consistent with the currently accepted standard of care in order to determine the comparative effectiveness of the two screening strategies. Participants will be surveyed annually to determine if they have undergone colonoscopy or been diagnosed with CRC.

The primary study endpoint will be CRC mortality within 10 years of enrollment. The secondary endpoints are (1) the incidence of CRC within 10 years of enrollment and (2) major complications of colonoscopy. Mortality will be determined through queries of the VA Vital Status File. Cause of death will be determined primarily using death certificates from the National Death Index-Plus database, augmented by adjudication of medical records for known CRC cases where CRC is not listed as a cause of death on the death certificate. The investigators postulate that screening colonoscopy will result in a 40% reduction in CRC mortality over 10 years relative to annual FIT screening. Using a log-rank test with a 2-sided test of significance, =0.05, a sample size of 50,000 participants will be required to test the primary hypothesis with 82% power, assuming a 1% annual rate of crossover from FIT to colonoscopy and a 0.5% annual rate of loss to follow-up. The planned study duration is 12.5 years with 2.5 years of recruitment and 10 years of follow-up for all enrolled participants.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged 50-75 years of age
* Veteran
* Able to provide informed consent

Exclusion Criteria:

* Symptoms of lower gastrointestinal tract disease warranting colonoscopic evaluation, including:

  * More than one episode of rectal bleeding within the past 6 months
  * Documented iron deficiency anemia
  * Significant documented unintentional weight loss (>10% of baseline weight) over 6 months
* Family history of CRC in a first degree relative at any age
* Prior history of colonic disease including:

  * Inflammatory bowel disease (e.g. ulcerative colitis or Crohn's disease)
  * One or more colorectal neoplastic polyps (i.e. adenomas)
  * Colorectal cancer
* Prior history of colonic resection
* Prior colonic examination, including:

  * Colonoscopy within the past 9.5 years
  * Sigmoidoscopy within the past 5 years
  * Barium enema within the past 5 years
  * CT colonography within the past 5 years
* gFOBT or FIT in the past 10 months
* Stool DNA test within the past 3 years
* Pregnancy
* Prisoner
* Significant comorbidity that would preclude benefit from screening or pose significant risk for the performance of colonoscopy (e.g. severe lung disease, end-stage renal disease, end-stage liver disease, severe heart failure, recent diagnosis of cancer (with the exception of non-melanoma skin cancer))
* Participation in a concurrent interventional study pertaining to the colon or rectum (including studies of colonoscopy or colorectal cancer screening. Waivers to this exclusion criteria can be requested and granted with the approval of the CONFIRM study co-chairs, the Cooperative Study Program and the leadership of the other study.
* Likely inability to track the individual over time (e.g. no permanent address at the time of screening for study entry)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50126 (Actual)
Dates: Start 2012-04-30 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is colorectal cancer mortality. | 10 years
  The primary outcome is colorectal cancer mortality. Patient survival will be monitored for 10 years, with survival assessed by both annual surveys and data reported to vital status registries, including the VA Vital Status File, which is comprised of the VA Beneficiary Identification and Records Locator System (BIRLS), the Medical SAS Inpatient Data Sets, and the Social Security Administration's Death Master File. The National Center for Health Statistics' National Death Index database will be used to find cause of death.

SECONDARY OUTCOMES:
FIT Positive - If Colonoscopy is Warranted | 10 Years
  There are no physical risks associated with performance of FIT screening. However, those with a positive FIT will be referred for evaluation by their primary care provider or site principal investigator to determine if colonoscopy is warranted. Those subsequently referred for colonoscopy will be exposed to its risks, and complications will be tracked as a secondary outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Jason A. Dominitz, MD MHS, Study Chair — VA Puget Sound Health Care System Seattle Division, Seattle, WA; Douglas J Robertson, MD MPH, Study Chair — White River Junction VA Medical Center, White River Junction, VT
Locations (46):
- United States (45):
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - Central Arkansas VHS John L. McClellan Memorial Veterans Hospital, Little Rock, AR, Little Rock, Arkansas
  - VA Central California Health Care System, Fresno, CA, Fresno, California
  - VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - Orlando VA Medical Center, Orlando, FL, Orlando, Florida
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - VA Pacific Islands Health Care System, Honolulu, HI, Honolulu, Hawaii
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - Robley Rex VA Medical Center, Louisville, KY, Louisville, Kentucky
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Kansas City VA Medical Center, Kansas City, MO, Kansas City, Missouri
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri
  - Manchester VA Medical Center, Manchester, NH, Manchester, New Hampshire
  - East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ, East Orange, New Jersey
  - Northport VA Medical Center, Northport, NY, Northport, New York
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Salisbury W.G. (Bill) Hefner VA Medical Center, Salisbury, NC, Salisbury, North Carolina
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Oklahoma City VA Medical Center, Oklahoma City, OK, Oklahoma City, Oklahoma
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Philadelphia MultiService Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island
  - Memphis VA Medical Center, Memphis, TN, Memphis, Tennessee
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - White River Junction VA Medical Center and Regional Office, White River Junction, VT, White River Junction, Vermont
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington
  - Clarksburg Louis A. Johnson VA Medical Center, Clarksburg, WV, Clarksburg, West Virginia
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin
- VA Caribbean Healthcare System, San Juan, PR, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dominitz JA, Robertson DJ, Ahnen DJ, Allison JE, Antonelli M, Boardman KD, Ciarleglio M, Del Curto BJ, Huang GD, Imperiale TF, Larson MF, Lieberman D, O'Connor T, O'Leary TJ, Peduzzi P, Provenzale D, Shaukat A, Sultan S, Voorhees A, Wallace R, Guarino PD. Colonoscopy vs. Fecal Immunochemical Test in Reducing Mortality From Colorectal Cancer (CONFIRM): Rationale for Study Design. Am J Gastroenterol. 2017 Nov;112(11):1736-1746. doi: 10.1038/ajg.2017.286. Epub 2017 Oct 10. PMID 29016565
- [Result] Robertson DJ, Dominitz JA, Beed A, Boardman KD, Del Curto BJ, Guarino PD, Imperiale TF, LaCasse A, Larson MF, Gupta S, Lieberman D, Planeta B, Shaukat A, Sultan S, Menees SB, Saini SD, Schoenfeld P, Goebel S, von Rosenvinge EC, Baffy G, Halasz I, Pedrosa MC, Kahng LS, Cassim R, Greer KB, Kinnard MF, Bhatt DB, Dunbar KB, Harford WV Jr, Mengshol JA, Olson JE, Patel SG, Antaki F, Fisher DA, Sullivan BA, Lenza C, Prajapati DN, Wong H, Beyth R, Lieb JG 2nd, Manlolo J, Ona FV, Cole RA, Khalaf N, Kahi CJ, Kohli DR, Rai T, Sharma P, Anastasiou J, Hagedorn C, Fernando RS, Jackson CS, Jamal MM, Lee RH, Merchant F, May FP, Pisegna JR, Omer E, Parajuli D, Said A, Nguyen TD, Tombazzi CR, Feldman PA, Jacob L, Koppelman RN, Lehenbauer KP, Desai DS, Madhoun MF, Tierney WM, Ho MQ, Hockman HJ, Lopez C, Carter Paulson E, Tobi M, Pinillos HL, Young M, Ho NC, Mascarenhas R, Promrat K, Mutha PR, Pandak WM Jr, Shah T, Schubert M, Pancotto FS, Gawron AJ, Underwood AE, Ho SB, Magno-Pagatzaurtundua P, Toro DH, Beymer CH, Kaz AM, Elwing J, Gill JA, Goldsmith SF, Yao MD, Protiva P, Pohl H, Kyriakides T; CONFIRM Study Group. Baseline Features and Reasons for Nonparticipation in the Colonoscopy Versus Fecal Immunochemical Test in Reducing Mortality From Colorectal Cancer (CONFIRM) Study, a Colorectal Cancer Screening Trial. JAMA Netw Open. 2023 Jul 3;6(7):e2321730. doi: 10.1001/jamanetworkopen.2023.21730. PMID 37432690
- [Derived] Shaukat A, Kahi CJ, Burke CA, Rabeneck L, Sauer BG, Rex DK. ACG Clinical Guidelines: Colorectal Cancer Screening 2021. Am J Gastroenterol. 2021 Mar 1;116(3):458-479. doi: 10.14309/ajg.0000000000001122. PMID 33657038